CLINICAL TRIAL: NCT02631551
Title: A Double-Blind, Randomized, Parallel-Group, Comparative Study to Evaluate the Efficacy, Safety and Tolerability of a Fixed Dose Combination GSP 301 Nasal Spray (NS) Compared With Placebo Nasal Spray and Individual Monotherapy Formulations (Comparators) in Subjects (Aged 12 Years and Older) With Seasonal Allergic Rhinitis (SAR)
Brief Title: Efficacy and Safety of Fixed Dose Combination GSP 301 Nasal Spray (NS) in the Treatment of Seasonal Allergic Rhinitis (SAR)
Acronym: GSP 301-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPL/CT/2014/016/III
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- GSP 301 NS (Experimental)
  Interventions: Drug: GSP 301 NS
- Olopatadine HCl NS (Active Comparator)
  Interventions: Drug: Olopatadine HCl NS
- Mometasone furoate NS (Active Comparator)
  Interventions: Drug: Mometasone furoate NS
- GSP 301 Placebo NS (Placebo Comparator)
  Interventions: Drug: GSP 301 Placebo NS

INTERVENTIONS:
Drug: GSP 301 NS — FDC of olopatadine HCl and mometasone furoate: 2 sprays in each nostril twice daily for 14 days
  Arms: GSP 301 NS
Drug: Olopatadine HCl NS — 2 sprays in each nostril twice daily for 14 days
  Arms: Olopatadine HCl NS
Drug: Mometasone furoate NS — 2 sprays in each nostril twice daily for 14 days
  Arms: Mometasone furoate NS
Drug: GSP 301 Placebo NS — 2 sprays in each nostril twice daily for 14 days
  Arms: GSP 301 Placebo NS

SUMMARY:
Study to evaluate the efficacy and safety of GSP 301 NS compared to placebo NS and to individual monotherapies (comparators) as well as the efficacy of these monotherapies (comparators) versus placebo NS over 14 days of study treatment

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 years and older inclusive of either sex.
2. Documented clinical history of SAR (for at least 2 years preceding the Screening Visit [Visit 1]) with exacerbations (clinical evidence of active symptoms) during the spring allergy season (tree/grass pollen)
3. A 12-hour reflective TNSS ≥ 8 out of a possible 12 and a congestion score of ≥ 2 for the AM assessment at the Screening Visit (Visit 1).

Exclusion Criteria:

1. Pregnant or lactating women.
2. Plans to travel outside the known pollen area for the investigative site for > 24 hours during the last 7 days of run in period.
3. History of anaphylaxis and/or other severe local reaction(s) to skin testing.
4. History of positive test for HIV, Hepatitis B or Hepatitis C infection.
5. Documented evidence of acute or significant chronic sinusitis or chronic purulent postnasal drip.
6. Subjects with an active pulmonary disorder or infection.
7. Subjects with posterior subcapsular cataracts or glaucoma

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, PhD, Study Director — Glenmark Pharmaceuticals
Locations (37):
- United States (37):
  - Investigational Site 20, Mission Viejo, California
  - Investigational Site 31, San Diego, California
  - Investigational Site 29, San Jose, California
  - Investigational Site 25, Centennial, Colorado
  - Investigational Site 22, Colorado Springs, Colorado
  - Investigational Site 10, Jupiter, Florida
  - Investigational Site 30, Miami, Florida
  - Investigational Site 37, Marietta, Georgia
  - Investigational Site 15, Stockbridge, Georgia
  - Investigational Site 23, Stockbridge, Georgia
  - Investigational Site 11, Louisville, Kentucky
  - Investigational Site 14, Baltimore, Maryland
  - Investigational Site 33, Wheaton, Maryland
  - Investigational Site 26, Ypsilanti, Michigan
  - Investigational Site 19, Minneapolis, Minnesota
  - Investigational Site 21, St Louis, Missouri
  - Investigational Site 16, Bellevue, Nebraska
  - Investigational Site 12, Skillman, New Jersey
  - Investigational Site 36, Rochester, New York
  - Investigational Site 18, Raleigh, North Carolina
  - Investigational Site 27, Cincinnati, Ohio
  - Investigational Site 34, Middleburg Heights, Ohio
  - Investigational Site 32, Medford, Oregon
  - Investigational Site 35, Portland, Oregon
  - Investigational Site 13, Orangeburg, South Carolina
  - Investigational Site 17, Spartanburg, South Carolina
  - Investigational Site 3, Austin, Texas
  - Investigational Site 5, Austin, Texas
  - Investigational Site 8, Austin, Texas
  - Investigational Site 1, Kerrville, Texas
  - Investigational Site 7, New Braunfels, Texas
  - Investigational Site 2, San Antonio, Texas
  - Investigational Site 4, San Antonio, Texas
  - Investigational Site 6, San Antonio, Texas
  - Investigational Site 9, San Antonio, Texas
  - Investigational Site 28, Waco, Texas
  - Investigational Site 24, Draper, Utah

REFERENCES:
- [Derived] Hampel FC, Pedinoff AJ, Jacobs RL, Caracta CF, Tantry SK. Olopatadine-mometasone combination nasal spray: Evaluation of efficacy and safety in patients with seasonal allergic rhinitis. Allergy Asthma Proc. 2019 Jul 3;40(4):261-272. doi: 10.2500/aap.2019.40.4223. Epub 2019 May 3. PMID 31053180

RESULTS

PARTICIPANT FLOW:
Groups:
- GSP 301 NS; Olopatadine HCl NS; Mometasone Furoate NS; GSP 301 Placebo NS: 2 sprays in each nostril twice daily for 14 days
Period: Overall Study
Arm/Group | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS | GSP 301 Placebo NS
Started | 302 | 297 | 294 | 287
Completed | 289 | 278 | 283 | 276
Not Completed | 13 | 19 | 11 | 11
Not completed — Adverse Event | 1 | 2 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 5
Not completed — Protocol deviation | 3 | 6 | 3 | 0
Not completed — Non-compliance with study procedures | 0 | 0 | 1 | 1
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0
Not completed — Other, specific reasons not collected | 5 | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS | GSP 301 Placebo NS | Total
Number analyzed (Participants) | 302 | 297 | 294 | 287 | 1180
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (15.4) | 39.6 (14.9) | 38.7 (16.3) | 39.4 (14.8) | 39.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 181 | 198 | 182 | 762
  Male | 101 | 116 | 96 | 105 | 418
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 0 | 3
  Asian | 2 | 4 | 7 | 7 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 1 | 4
  Black or African American | 56 | 67 | 59 | 48 | 230
  White | 241 | 219 | 224 | 231 | 915
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 3 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Average AM and PM Subject-reported 12-hour Reflective Total Nasal Symptoms Score (rTNSS) From Baseline to End of Treatment.
Description: Reflective Total Nasal Symptom Score (rTNSS) was calculated as the sum of 12-hour reflective scoring of the severity of four nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing). Subjects responded on a 4-point severity scale with scores ranging from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Time Frame: 14 days
Population: The Full Analysis Set (FAS) was defined as all subjects who were randomized and received at least one dose of investigational product and had at least one post-baseline primary efficacy assessment. This was the primary analysis set for efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS | GSP 301 Placebo NS
Number analyzed (Participants) | 299 | 294 | 294 | 283
units on a scale
  Baseline | 10.1 (1.2) | 10.3 (1.3) | 10.2 (1.2) | 10.2 (1.2)
  Change from baseline to end of treatment | -3.6 (3.2) | -3.2 (3.1) | -3.5 (3.3) | -2.8 (3.2)
Statistical Analysis 1: Comparison: GSP 301 NS vs GSP 301 Placebo NS; GSP 301 NS vs GSP 301 placebo NS comparison for rTNSS was tested at 0.05 significance level; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: GSP 301 NS vs Olopatadine HCl NS; GSP 301 NS vs Olopatadine HCl NS comparison for rTNSS was tested at 0.05 significance level; Test type: Superiority; p = 0.0029, Mixed Models Analysis
Statistical Analysis 3: Comparison: GSP 301 NS vs Mometasone Furoate NS; GSP 301 NS vs Mometasone furoate NS comparison for rTNSS was tested at 0.05 significance level; Test type: Superiority; p = 0.0587, Mixed Models Analysis
Statistical Analysis 4: Comparison: Olopatadine HCl NS vs GSP 301 Placebo NS; Olopatadine HCl NS vs GSP 301 Placebo NS comparison for rTNSS was tested at 0.05 significance level; Test type: Superiority; p = 0.0755, Mixed Models Analysis
Statistical Analysis 5: Comparison: Mometasone Furoate NS vs GSP 301 Placebo NS; Mometasone furoate NS vs GSP 301 Placebo NS comparison for rTNSS was tested at 0.05 significance level; Test type: Superiority; p = 0.0043, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The AEs and SAEs were collected from the time of signing the informed consent form until the end of study i.e., screening visit followed by 7-10 days of placebo run-in period and 14 days of treatment.
Arm/Group | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS | GSP 301 Placebo NS
All-Cause Mortality (participants affected / at risk) | 0/302 | 0/297 | 0/294 | 0/287
Serious Adverse Events (participants affected / at risk) | 1/302 | 0/297 | 0/294 | 0/287
Other Adverse Events (participants affected / at risk) | 0/302 | 0/297 | 0/294 | 0/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 NS (N=302) | Olopatadine HCl NS (N=297) | Mometasone Furoate NS (N=294) | GSP 301 Placebo NS (N=287)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the agreement, Sponsor reserves the right for publishing trial results and the Investigator cannot publish without written consent from the CRO/Sponsor.